CLINICAL TRIAL: NCT03010865
Title: Sodium Butyrate As A Treatment For Improving Cognitive Function In Schizophrenia
Brief Title: Sodium Butyrate For Improving Cognitive Function In Schizophrenia
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: sponsor withdrew the funds because the smell of sodium butyrate made blinding impossible
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016-12
Record Dates: First submitted 2016-12-28; First posted 2017-01-05 (Estimated); Last update posted 2019-01-17 (Actual); Status verified 2017-06

CONDITIONS: Schizophrenic Disorder; Cognitive Impairment
Keywords: HDAC inhibitors; Inflammation
MeSH Terms: conditions — Schizophrenia; Cognitive Dysfunction; Inflammation | interventions — Butyric Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sodium Butyrate (Experimental): Dietary Supplement: Sodium Butyrate 4.38 gms of sodium butyrate per day for 12 weeks
  Interventions: Drug: Sodium Butyrate
- Placebo Oral Capsule (Placebo Comparator): Placebo Oral Capsule placebo capsules containing approximately 9 mg of sodium butyrate per day
  Interventions: Drug: Placebo Oral Capsule

INTERVENTIONS:
Drug: Sodium Butyrate — Sodium butyrate is being supplied by T.E. Neesby (Brain White, T.E. Neesby, Inc.) in 730 mg capsules. The company asserts that their material is 98% pure and food grade. We will have identical placebo capsules. Subjects will receive 3 capsules twice daily (morning and late afternoon or evening) for a total of 4380 mg/day.
  Arms: Sodium Butyrate
Drug: Placebo Oral Capsule — Placebo Oral Capsule is also being supplied by T.E. Neesby (Brain White, T.E. Neesby, Inc.) and there is no difference from appearance, smell and taste. It contains 1.5 mg sodium butyrate per capsule. Subjects will receive 3 capsules twice daily (morning and late afternoon or evening) for a total of 9 mg/day.
  Arms: Placebo Oral Capsule

SUMMARY:
The purpose of this grant is to evaluate the efficacy of sodium butyrate as a novel treatment for cognitive deficits in schizophrenia (SZ). The aims will be to evaluate its effects on improving symptoms and functioning in SZ, and the relationship of the drug's clinical effects to epigenetic and inflammation related biochemical changes.

DETAILED DESCRIPTION:
The persistent cognitive deficits which can be appreciated across the course of SZ, from prodromal to chronic SZ, may be the most important underlying dysfunction in preventing functional, occupational, and social recovery in SZ compared to other symptom domains. Sodium butyrate is a short chain fatty acid and binds to the zinc site of histone deacetylases (HDAC). The inhibition of HDAC results in histone hyperacetylation. This study aims to evaluate its effects on improving symptoms and functioning in SZ, and the relationship of the drug's clinical effects to epigenetic and inflammation related biochemical changes.

The proposed study will be a double blind study of the effects of sodium butyrate on cognitive function and symptoms in chronic SZ patients showing continued cognitive deficits.The primary specific aims of the proposal will be to test the the MATRICS (MCCB) battery,delayed recall performance, and performance on real world functional tasks as assessed by the USCD Performance- Based Skills Assessment Battery (UPSA). In addition, we will also investigate whether sodium butyrate may improve other aspects of cognition.

We will also explore whether improvement in cognition is related to change in HDAC activity in peripheral blood cells and changes in inflammatory makers in the blood, and assess whether there is any improvement in psychopathology as measured by PANSS scale.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have cognitive deficits as indicated by a score of < 85 on RBANS,
2. meet criteria for DSM-5 diagnosis of chronic SZ, schizoaffective disorder (SA),
3. Subjects who are stably treated with antipsychotic medications and are not in acute exacerbation of illness symptoms.

Exclusion Criteria:

1. History of mental retardation or pervasive developmental disorder,
2. Subjects with a current serious neurological/CNS disorder (such as seizure disorder, stroke or multiple sclerosis) or brain trauma,
3. Current treatment with valproic acid, butyrate drugs, sulforaphane, or other drugs or chemicals known to have high HDAC inhibitory activity,
4. Pregnancy,
5. Severe unstable medical condition,
6. Current suicidal or homicidal thoughts,
7. Current alcohol or substance abuse (other than nicotine or occasional marijuana) in the last month.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in MATRICS Battery Score | Basline, week 6, up to 12 weeks
  MATRICS Cognitive Battery

SECONDARY OUTCOMES:
Change from baseline in Logical Memory Test score | Basline, up to 12 weeks
  Logical Memory Test for longer term memory
Change from baseline in Positive and Negative Syndrome Scale (PANSS) total score | Basline, week 6, up to 12 weeks
  Positive and Negative Syndrome Scale (PANSS) symptom rating scale
Change from baseline in Paced Auditory Serial Addition Test (PASAT) score | Basline, week 6, up to 12 weeks
  Alternate working memory test
Change from baseline in UCSD Performance-Based Skills Assessment (UPSA) total score | Baseline, up to 12 weeks
  University of California, San Diego (UCSD) Performance-Based Skills Assessment Battery

OTHER OUTCOMES:
Change from baseline in Side-Effect Scale Score | Basline, week 2, week 6, up to 12 weeks
  Patient self-report of side-effects of active or placebo medication

CONTACTS AND LOCATIONS:
Overall Officials: Chunbo Li, M.D., Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Stanley foundation requests: Based on the terms of your award, Stanley Medical Research Institute (SMRI) now requires submission of the individual patient data from all SMRI funded studies. In order to make the process as efficient as possible and provide a secure location for study data, National Institute of Mental Health (NIMH) is graciously allowing SMRI access to their National Database for Clinical Trials (NDCT) to collect and house data.